CLINICAL TRIAL: NCT00432081
Title: Effect of Indomethacin on the Progression of Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: American Health Assistance Foundation (Other); Netherlands Brain Foundation (Other); Netherlands Alzheimer Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2001-15-DDJ; 917.46.331
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2007-02-06 (Estimated); Status verified 2007-02

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Inflammation; Anti-Inflammatory Agents; Anti-Inflammatory Agents, Non-Steroidal; Drug Therapy
MeSH Terms: conditions — Alzheimer Disease; Dementia; Inflammation | interventions — Indomethacin

INTERVENTIONS:
Drug: indomethacin

SUMMARY:
The purpose of this study is determine whether indomethacin is able to retard disease progression in patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Previous research indicates that inflammation plays a role in the pathogenesis of Alzheimer's disease (AD), and nonsteroidal anti-inflammatory drugs (NSAIDs) may retard the progression of the disease.

Comparison(s): Cognitive decline of patients with mild to moderate AD receiving the NSAID indomethacin, compared to cognitive decline of patients with mild to moderate AD receiving placebo, during a one-year period.

ELIGIBILITY:
Inclusion Criteria:

* The patient will satisfy the DSM-IV criteria for dementia of the Alzheimer's type.
* The patient will satisfy the NINCDS/ADRDA criteria for the clinical diagnosis of probable Alzheimer's disease (Appendix I).
* The severity of dementia for each patient will be quantified by a Mini-Mental State Examination (MMSE) score between 10 and 26 (both inclusive).
* The patient is living at home or in a home for the elderly.
* The patient has a responsible caregiver who is able to provide information about the patient's functional status.
* Written informed consent is obtained from the patient or the legally accepted representative.

Exclusion Criteria:

* The patient satisfies the NINDS-AIREN criteria for probable vascular dementia.
* A known exaggerated pharmacological sensitivity or allergy to NSAID's.
* History of peptic ulceration, gastric surgery or gastrointestinal bleeding.
* Current diagnosis of active peptic ulceration.
* Current diagnosis of severe and unstable cardiovascular disease.
* Current diagnosis of renal failure.
* Advanced, severe and unstable disease of any type, other than Alzheimer's disease, that may interfere with primary and secondary variable evaluations, including a medical condition which should be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical or mental status of the patient to a significant degree or put the patient at special risk.
* Intake of any of the following concomitant medications: salicylates, coumarin derivatives, ACE-inhibitors, loop diuretics.
* Intake of any of the following concomitant medications more than two months immediately prior or during the study: NSAID's, systemic corticosteroids.
* Intake of any of the following concomitant medications with a possible effect on cognition: estrogen, deprenyl, vitamin E, neuroleptics, anticholinergics. Patients using stable doses of cholinesterase inhibitors were eligible, with the provision that the dose should not be changed during the study. Cholinesterase inhibitors could not be initiated during the study.
* Excessive use of alcohol (more than 5 units per day)
* The patient is, either alone or with the aid of a caregiver, not able to reliably take the medication.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2000-05; Study Completion 2005-08

PRIMARY OUTCOMES:
Score on the Cognitive subscale of the Alzheimer's Disease Assessment Scale at 12 months.

SECONDARY OUTCOMES:
Score on the Noncognitive subscale of the Alzheimer's Disease Assessment Scale at 12 months
Score on the Clinician Interview-Based Impression of Change with caregiver input at 12 months
Score on the Mini-Mental State Examination at 12 months
Score on the Neuropsychiatric Inventory at 12 months
Score on the The Interview for Deterioration in Daily living activities in Dementia at 12 months
The occurrence of adverse events during 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rene WM Jansen, MD, PhD, Principal Investigator — Radboud University Medical Center Nijmegen; Berry PH Kremer, MD, PhD, Principal Investigator — Radboud University Medical Center Nijmegen; Danielle De Jong, MD, Study Director — Radboud University Medical Center Nijmegen
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem
  - Radboud University Medical Center, Nijmegen

REFERENCES:
- [Background] Rogers J, Kirby LC, Hempelman SR, Berry DL, McGeer PL, Kaszniak AW, Zalinski J, Cofield M, Mansukhani L, Willson P, et al. Clinical trial of indomethacin in Alzheimer's disease. Neurology. 1993 Aug;43(8):1609-11. doi: 10.1212/wnl.43.8.1609. PMID 8351023
- [Background] McGeer PL, McGeer EG. NSAIDs and Alzheimer disease: epidemiological, animal model and clinical studies. Neurobiol Aging. 2007 May;28(5):639-47. doi: 10.1016/j.neurobiolaging.2006.03.013. Epub 2006 May 11. PMID 16697488
- [Derived] de Jong D, Jansen R, Hoefnagels W, Jellesma-Eggenkamp M, Verbeek M, Borm G, Kremer B. No effect of one-year treatment with indomethacin on Alzheimer's disease progression: a randomized controlled trial. PLoS One. 2008 Jan 23;3(1):e1475. doi: 10.1371/journal.pone.0001475. PMID 18213383